CLINICAL TRIAL: NCT03108560
Title: A Multi-center, Randomized-controlled, Open-label Clinical Trial: Sublobar Resection Versus Lobectomy for cT1N0M0 Non-small-cell Lung Cancer
Brief Title: Sublobar Resection Versus Lobectomy for cT1N0M0 Non-small-cell Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Ruijin Hospital (Other); RenJi Hospital (Other); Fujian Medical University Union Hospital (Other); The Second Affiliated Hospital of Dalian Medical University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Ningbo No.2 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZSTS201701
Record Dates: First submitted 2017-03-28; First posted 2017-04-11 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: sublobar resection; lobectomy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Anterior Temporal Lobectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sublobar group (Experimental): Patients receive sublobar resection, including wedge resection and segmentectomy.
  Interventions: Procedure: sublobar resection
- Lobectomy group (Active Comparator): Patients receive lobectomy.
  Interventions: Procedure: lobectomy

INTERVENTIONS:
Procedure: sublobar resection — Patients receive sublobar resection, which includes wedge resection and segmentectomy.
  Arms: Sublobar group
Procedure: lobectomy — patients receive lobectomy
  Arms: Lobectomy group

SUMMARY:
The incidence rate of ground-glass opacity (GGO) has been increasing these years. A great number of retrospective studies suggested that sublobar resection was better for some GGO patients. However, no prospective clinical study supports the perspective. This study is prospective, multi-center, randomized-controlled. The aim of this study is to investigate whether sublobar resection is inferior to lobectomy for cT1N0M0 non-small-cell lung cancer or not.

ELIGIBILITY:
Inclusion Criteria:

* cT1N0M0 non-small-cell lung cancer
* ground-glass opacity, ≤2cm, GGO≥25%
* eligible for both lobectomy and sublobar resection
* intraoperative pathology is minimally-invasive adenocarcinoma or invasive adenocarcinoma
* intraoperative pathology of biopsied station 10 lymph node is negative

Exclusion Criteria:

* intraoperative pathology is benign nodule, atypical adenomatous hyperplasia, or adenocarcinoma in-situ
* intraoperative pathology of biopsied station 10 lymph node is positive
* multiple GGOs, lesions other than dominant lesion are malignant or >5mm
* history of thoracic surgery
* history of malignancy in recent 5 years
* unstable systemic disease
* patients with psychiatric disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2017-04-18 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | five years after surgery
  survival status of patients after surgery

SECONDARY OUTCOMES:
Disease Free Survival | five years after surgery
  recurrence status of patients after surgery
Local and distant recurrence rates | five years after surgery
  recurrence rate of local and distant locations respectively
Pulmonary Function: forced expiratory volume in 1 second (FEV1) in liter | 3rd, 6th, 12th, and 24th month after surgery
  FEV1 of patients after surgery
Pulmonary Function: forced vital capacity (FVC) in liter | 3rd, 6th, 12th, and 24th month after surgery
  FVC of patients after surgery
Pulmonary Function: diffusing capacity of the lungs for carbon monoxide (DLCO) in mL/min/mmHg | 3rd, 6th, 12th, and 24th month after surgery
  DLCO of patients after surgery
Morbidity rate | up to 30 days after surgery
  the rates of complications related to treatment during perioperative period
Mortality rate | up to 30 days after surgery
  the rates of death related to treatment during perioperative period

CONTACTS AND LOCATIONS:
Overall Officials: Di Ge, MD, Study Chair — Fudan University
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The data of all case report forms are to be collected and shared with other researchers at the end of followup.